CLINICAL TRIAL: NCT02232802
Title: Comparative, Randomized, Single-dose, 2-way Cross Over Bioavailability Study of Enoxaparin Sodium Chemi (80 mg/0.8mL) and Clexane® (80 mg/0.8mL) s.c. in Healthy Adult Subjects Under Fasting Conditions.
Brief Title: Bioavailability Study of Enoxaparin Sodium Chemi and Clexane s.c.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chemi S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: ENOXA/14/2
Record Dates: First submitted 2014-09-03; First posted 2014-09-05 (Estimated); Results first posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Enoxaparin Sodium is Administered to Healthy Volunteers
MeSH Terms: interventions — enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin Sodium Chemi (Experimental): Enoxaparin Sodium Chemi and Clexane will be administered to healthy subjects. Each subject will receive each treatment over two separate treatment periods under fasting conditions.
  Interventions: Drug: Enoxaparin Sodium
- Clexane (Experimental): Enoxaparin Sodium Chemi and Clexane will be administered to healthy subjects. Each subject will receive each treatment over two separate treatment periods under fasting conditions.
  Interventions: Drug: Enoxaparin Sodium

INTERVENTIONS:
Drug: Enoxaparin Sodium — comparison of bioavailability of generic Enoxaparin Sodium and Clexane
  Other Names: Clexane
  Arms: Enoxaparin Sodium Chemi
Drug: Enoxaparin Sodium — comparison of bioavailability of generic Enoxaparin Sodium and Clexane
  Other Names: generic Enoxaparin Sodium
  Arms: Clexane

SUMMARY:
* The primary objective of the trial is to assess the single-dose relative bioavailability of Chemi Enoxaparin (80 mg/0.8 mL) and Clexane® (80 mg/0.8 mL) administered by subcutaneous (s.c.) injection, under fasting conditions in healthy volunteers.
* The secondary objective of the trial is to assess safety and tolerability of Chemi Enoxaparin (80 mg/0.8 mL) and Clexane® (80 mg/0.8 mL) administered by s.c. injection, under fasting conditions in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, randomised, single-dose, 2-way crossover study to determine the comparative bioavailability of enoxaparin sodium from the Chemi Enoxaparin s.c. (80 mg/0.8mL) with that from the reference IMP, Clexane® s.c. (80 mg/0.8mL), following single dose administration in healthy male and female subjects.

Each subject received each treatment over two separate treatment periods under fasting conditions. Each dosing day for male subjects will be separated by a washout period of at least 7 days. The study comprised a pre-study screen (within 14 days of the first dose), followed by 2 Treatment Periods (1 and 2). During each treatment period, subjects will reside at Simbec from the evening before dosing (Day 1), until at least 36 h post dose (evening of Day 2). On admission (Day -1), subjects will provide a urine sample for a drugs of abuse screen; this sample will also be tested to confirm a negative pregnancy result in female volunteers.

A single dose of the randomised treatment will be given on the morning of Day 1 following an overnight fast and blood PK/PD samples collected from pre-dose up to 36 h post dose (14 samples). Safety will also be evaluated at specified times throughout the study.

The post study visit will be conducted on Day 2 (36 h post-dose) of Treatment Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female volunteer between 18 and 55 years of age.
* Subject with a BMI of 18-30 (Body Mass Index = Body weight (kg) / [Height (m)]2)
* Subject with no clinically significant abnormal serum biochemistry, haematology, coagulation factors and urine examination values within 14 days of the first dose.
* Subject with no clinically significant abnormalities in 12-lead electrocardiogram (ECG) and vital signs determined within 14 days of the first dose.
* Subject with negative human immunodeficiency virus (HIV) and hepatitis B surface antigen (HbsAg) and hepatitis C virus antibody (HCV) results.

Exclusion Criteria:

* Subject with hypersensitivity or idiosyncratic reaction to enoxaparin and/or low molecular weight heparins, and/or pork products.
* Subject with a relevant history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease. Or with history or presence of alcoholism or drug abuse;
* Subject with clinically relevant abnormal physical findings or clinically relevant abnormal laboratory values indicative of physical illness;
* Female subject who is pregnant or lactating
* Female subject with weight < 45 kg or male subject with weight < 57 kg.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2014-12-05 (Actual); Study Completion 2014-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bettica, MD, Study Director — Italfarmaco S.p.A.
Locations (1):
- Simbec Research Ltd, Merthyr Tydfil, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-seven (47) subjects (23 male and 24 female) were enrolled in the study. The subjects were selected from a large panel who offered their services as healthy volunteers for the purpose of undertaking REC and Regulatory Authority-approved studies on drug safety, absorption and disposition.
Pre-assignment Details: The study comprised a screening visit and 2 treatment periods. Only two doses were scheduled to be administered: first dose (period 1) - wash out (at least 7 days) - 2nd dose (period 2) - wash out period (at least 7 days). Each treatment period was of 2 days duration. Screening assessments: from Day -14 to Day -1.
Groups:
- Test IMP - Reference IMP: These patients reveiced the following sequence:
  Test IMP: A single-dose of 80mg/0.8 mL Chemi Enoxaparin. Reference IMP: A single-dose of 80mg/0.8 mL Clexane® Each dose was administered s.c. into the left or right side of the abdomen (alternating sides with treatment period).
  Each dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti-FXa activity) in 0.8 mL water for injection.
  Subjects remained in an upright position whilst receiving each dose and for 4 h afterwards.
  There were at least 7 days between each dose administration for males and female subjects of nonchildbearing potential. Female subjects of child bearing potential underwent a washout period of approximately 28 days.
- Reference IMP - Test IMP: These patients reveiced the following sequence:
  Reference IMP: A single-dose of 80mg/0.8 mL Clexane® Test IMP: A single-dose of 80mg/0.8 mL Chemi Enoxaparin. Each dose was administered s.c. into the left or right side of the abdomen (alternating sides with treatment period).
  Each dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti-FXa activity) in 0.8 mL water for injection.
  Subjects remained in an upright position whilst receiving each dose and for 4 h afterwards.
  There were at least 7 days between each dose administration for males and female subjects of nonchildbearing potential.
  Female subjects of child bearing potential underwent a washout period of approximately 28 days.
Period: Period 1
Arm/Group | Test IMP - Reference IMP | Reference IMP - Test IMP
Started | 24 | 23
Completed | 22 | 22
Not Completed | 2 | 1
Not completed — Sponsor request | 1 | 0
Not completed — Adverse Event | 1 | 1
Period: Washout
Arm/Group | Test IMP - Reference IMP | Reference IMP - Test IMP
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Test IMP - Reference IMP | Reference IMP - Test IMP
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0
Period: Washout
Arm/Group | Test IMP - Reference IMP | Reference IMP - Test IMP
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test IMP - Reference IMP | Reference IMP - Test IMP | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 23 | 47
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 11 | 12 | 23
Region of Enrollment [Number; unit: participants]
  United Kingdom | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Anti-FXa and Anti-FIIa)
Description: Cmax is the maximum measured plasma activity/concentration. Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: PK population: All subjects who received study medication in both treatment periods, had sufficient plasma activity/concentration-time profiles and who did not violate the protocol in such a way that may have invalidated or biased the results (major protocol violators) were included in the PK analysis.
Measure: Mean (Standard Deviation); unit: IU/mL
Groups:
- Enoxaparin Sodium Chemi (Test IMP): Enoxaparin Sodium Chemi (i.e. Test IMP) was administered to healthy subjects. A single dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti-FXa activity) in 0.8 mL water for injection. It was administered s.c . into the right or left side of the abdomen (alternating sides with treatment period).
- Clexane (Reference IMP): Clexane (i.e. Reference IMP) was administered to healthy subjects. A single dose contained 80 mg enoxaparin sodium (equivalent to 8,000 international units (IU) anti-factor Xa (anti-FXa activity) in 0.8 mL water for injection. It was administered s.c . into the right or left side of the abdomen (alternating sides with treatment period).
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
IU/mL
  Anti-FXa | 0.8593 (0.18056) | 0.8698 (0.20921)
  Anti-thrombin/factor IIa | 0.1187 (0.03451) | 0.1296 (0.03713)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Statistical comparison for Anti-FXa; Test type: Equivalence — Following logarithmic transformation, Cmax values were subjected to an analysis of variance (ANOVA), including fixed effects for sequence, period, treatment and subject nested within sequence; least square mean difference ratio = 99.42, 95% CI 2-sided [96.28 to 102.65] — Geometric least square means are being compared
Statistical Analysis 2: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Statistical comparison on Anti-FIIa; Test type: Equivalence — Following logarithmic transformation, Cmax was subjected to an analysis of variance (ANOVA), including fixed effects for sequence, period, treatment and subject nested within sequence; least square mean difference ratio = 91.55, 95% CI 2-sided [86.65 to 96.73] — Geometric least square means are being compared

2. Primary Outcome: AUC0-t (Anti-FXa and Anti-FIIa)
Description: AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method. Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII). thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa).
  As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
h*IU/mL
  Anti-FXa | 9.6259 (1.68590) | 9.3927 (1.83943)
  Anti-FIIa | 1.0234 (0.28817) | 1.1097 (0.31668)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FXa statistical comparison; Test type: Equivalence — Following logarithmic transformation, AUC0-t values were subjected to an analysis of variance (ANOVA), including fixed effects for sequence, period, treatment and subject nested within sequence; least square mean difference ratio = 102.89, 95% CI 2-sided [100.67 to 105.15] — Geometric least square means are being compared
Statistical Analysis 2: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FIIa comparison; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; least square mean difference ratio = 92.37, 95% CI 2-sided [87.72 to 97.25] — Geometric least square means are being compared

3. Secondary Outcome: AUC0-inf (Anti-FXa and Anti-FIIa)
Description: AUC0-inf is the area under the activity/concentration-time curve from time 0 extrapolated to infinity. It was calculated as the sum of AUC0-t plus the ratio of the last measurable value to the elimination rate constant. Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 43
h*IU/mL
  Anti-FXa | 10.2789 (1.71377) | 9.9197 (1.86143)
  Anti-FIIa: number analyzed (Participants) | 36 | 39
  Anti-FIIa | 1.1489 (0.29243) | 1.2926 (0.40401)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FXA comparison; Test type: Equivalence — Following logarithmic transformation, AUC0-inf values were subjected to an analysis of variance (ANOVA), including fixed effects for sequence, period, treatment and subject nested within sequence; least square mean ratio = 104.26, 95% CI 2-sided [101.68 to 106.9] — Geometric least square means are being compared
Statistical Analysis 2: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FIIa comparison; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; least square mean ratio = 90.44, 95% CI 2-sided [85.38 to 95.8] — Geometric least square means are being compared

4. Secondary Outcome: Tmax (Anti-FXa and Anti-FIIa)
Description: Tmax is the time to Cmax. Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
Hours
  Anti-FXa | 4.0000 [2.000 to 6.000] | 4.0000 [3.000 to 6.000]
  Anti-FIIa | 4.0000 [2.000 to 6.000] | 4.0000 [3.000 to 16.000]
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FXa comparison; Test type: Equivalence — An assessment of tmax was performed using the Wilcoxon matched pairs test. In addition, a 95 % non-parametric CI was constructed for the median difference in tmax based on the method of Campbell and Gardner; p = 0.7642, Wilcoxon (Mann-Whitney) — An assessment of tmax was performed using the Wilcoxon matched pairs test. In addition, a 95 % non-parametric CI was constructed for the median difference in tmax based on the method of Campbell and Gardner; least square mean ratio = 0, 95% CI 2-sided [-0.5 to 0.5] — Geometric least square means are being compared
Statistical Analysis 2: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Anti-FIIa comparison; Test type: Equivalence — [test comment as in outcome 4, analysis 1]; p = 0.9464, Wilcoxon (Mann-Whitney); least square mean ratio = 0, 95% CI 2-sided [-0.5 to 0.5] — Geometric least square means are being compared

5. Secondary Outcome: Lambda Zeta (Anti-FXa and Anti-FIIa)
Description: Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration vs time curve.
  Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 43
1/hour
  Anti-FXa | 0.0962 (0.04251) | 0.1133 (0.04337)
  Anti-IIa: number analyzed (Participants) | 36 | 39
  Anti-IIa | 0.2111 (0.10435) | 0.1938 (0.11612)

6. Secondary Outcome: t1/2 (Anti-FXa and Anti-FIIa)
Description: T1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 43
hours
  Anti-FXa | 8.4757 (3.22737) | 6.9507 (2.42567)
  Anti-FIIa: number analyzed (Participants) | 36 | 39
  Anti-FIIa | 4.6214 (2.97971) | 6.5045 (8.67539)

7. Secondary Outcome: Tmin (Anti-FXa and Anti-FIIa)
Description: Tmin is the time of Cmin. Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
hours
  Anti-FXa | 0.00 (0.000) | 0.00 (0.000)
  Anti-FIIa | 4.18 (8.538) | 6.91 (12.211)

8. Secondary Outcome: AUC%ex (Anti-FXa and Anti-FIIa)
Description: AUC%ex is the residual area, i.e. the percentage of the area under the curve (AUC) extrapolated to infinity observed from Tlast to infinity.
  Blood samples (2 x 10 mL) for determination of plasma anti-FIIa and anti-FXa were collected from a forearm vein into a Citrate Sarstedt Monovette at the following time-points (at day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)) and kept frozen until analysis.
  Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti-FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total value of AUC
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 43
percentage of total value of AUC
  Anti-FXa | 6.4515 (2.68130) | 4.9683 (1.80897)
  Anti-FIIa: number analyzed (Participants) | 36 | 39
  Anti-FIIa | 12.0593 (7.68842) | 12.0906 (9.02925)

9. Secondary Outcome: Cmin (Anti-FXa and Anti-FIIa)
Description: Cmin is the minimum plasma activity/concentration. Enoxaparin exerts its anti-coagulant effect primarily via interaction with anti-thrombin III (ATIII), thereby enhancing the inhibitory effect of ATIII on activated factor Xa (FXa) and thrombin/factor IIa (FIIa). As enoxaparin cannot be measured directly in blood, the PK of enoxaparin have been studied on the basis of its effect on clotting mechanisms, particularly the inhibition of FXa (anti-FXa) and FIIa (anti- FIIa) activity. Results are presented as derived plasma PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
IU/mL
  Anti-FXa | 0.000 (0.0000) | 0.000 (0.0000)
  Anti-FIIa | 0.002 (0.0044) | 0.002 (0.0042)

10. Secondary Outcome: Cmax (Tissue Factor Pathway Inhibitor, TFPI)
Description: Cmax is the maximum measured plasma activity/concentration. Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
IU/mL | 2.4327 (0.35998) | 2.3391 (0.33903)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — Results obtained using a fixed effects ANOVA with fixed effects for sequence, period, treatment and subject nested within sequence; Geometric least square mean ratio = 103.94, 95% CI 2-sided [101.22 to 106.73]

11. Secondary Outcome: Cmax (Anti-FXa/Anti-FIIa Ratio)
Description: Cmax is the maximum measured plasma activity/concentration. The ratio of anti-FXa/anti-FIIa activity was calculated for each parameter. Reults are presented as derived ratio of PK parameters.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
ratio | 7.4450 (1.04983) | 6.8546 (0.95651)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Geometric least square mean ratio = 108.59, 95% CI 2-sided [103.93 to 113.46]

12. Secondary Outcome: AUC0-t (Derived Thrombin Generation)
Description: AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
  Thrombin generated in the thrombin generation test can be quantified as platelet-rich or platelet-poor plasma using the calibrated automated thrombogram method, which monitors the cleavage of a fluorogenic substrate that is simultaneously compared to the known thrombin activity in a non-clotting plasma sample.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nM
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
h*nM | 3731.0710 (1375.97298) | 3597.3375 (1104.52084)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Geometric least square mean ratio = 102.76, 95% CI 2-sided [97.51 to 108.28]

13. Secondary Outcome: Cmin (Derived Thrombin Generation)
Description: Thrombin generated in the thrombin generation test can be quantified as platelet-rich or platelet-poor plasma using the calibrated automated thrombogram method, which monitors the cleavage of a fluorogenic substrate that is simultaneously compared to the known thrombin activity in a non-clotting plasma sample.
  Cmin is the minimum plasma activity/concentration.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
nM | 13.534 (7.6300) | 11.543 (6.9299)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Geometric least square mean ratio = 114.91, 95% CI 2-sided [102.29 to 129.08]

14. Secondary Outcome: Tmin (Derived Thrombin Generation)
Description: Thrombin generated in the thrombin generation test can be quantified as platelet-rich or platelet-poor plasma using the calibrated automated thrombogram method, which monitors the cleavage of a fluorogenic substrate that is simultaneously compared to the known thrombin activity in a non-clotting plasma sample. Tmin is the time of Cmin.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
hours | 3.67 (1.136) | 3.64 (0.911)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; p = 0.8554, ANOVA; Median Difference (Final Values) = 0, 95% CI 2-sided [-0.5 to 0.5]

15. Secondary Outcome: AUC0-t (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*Unit/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
h*Unit/mL | 56.1828 (7.91060) | 55.7851 (8.43154)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; geometric least square mean ratio = 100.86, 95% CI 2-sided [99.27 to 102.47]

16. Secondary Outcome: AUC0-inf (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  AUC0-inf is the area under the activity/concentration-time curve from time 0 extrapolated to infinity. It was calculated as the sum of AUC0-t plus the ratio of the last measurable value to the elimination rate constant.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*Unit/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 23 | 18
h*Unit/mL | 140.8383 (36.06655) | 173.9833 (123.89404)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; geometric least square mean ratio = 95.13, 95% CI 2-sided [85.7 to 105.6]

17. Secondary Outcome: Tmax (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  Tmax is the time to Cmax
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
hours | 1.7500 (0.83178) | 1.8068 (1.20665)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — An assessment of tmax was performed using the Wilcoxon matched pairs test. In addition, a 95 % nonparametric CI was constructed for the median difference in tmax based on the method of Campbell and Gardner; p = 0.6857, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.25 to 0.5] — Median difference is the difference between median tmax in Test IMP versus Reference IMP arms

18. Secondary Outcome: Cmin (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  Cmin is the minimum plasma activity/concentration.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Unit/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
Unit/mL | 1.261 (0.2277) | 1.290 (0.2288)

19. Secondary Outcome: Tmin (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  Tmin is the time of Cmin.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
hours | 16.27 (5.275) | 15.55 (6.293)

20. Secondary Outcome: T1/2 (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI), which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  T1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 23 | 18
hours | 41.6397 (8.66880) | 57.2439 (46.13993)

21. Secondary Outcome: Lambda Zeta (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also releases tissue factor pathway inhibitor (TFPI)[5], which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration vs time curve.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 23 | 18
1/hour | 0.0172 (0.00323) | 0.0148 (0.00440)

22. Secondary Outcome: AUC%ex (Tissue Factor Pathway Inhibitor, TFPI)
Description: Enoxaparin also release tissue factor pathway inhibitor (TFPI)[5], which is thought to contribute to anti-coagulant activity, by inhibiting FXa generation and free FXa.
  AUC%ex is the residual area, i.e. the percentage of the area under the curve (AUC) extrapolated to infinity observed from Tlast to infinity.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total AUC
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 23 | 18
percentage of total AUC | 58.9149 (5.07416) | 63.0497 (8.81000)

23. Secondary Outcome: AUC0-t (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  AUC0-t is the area under the plasma activity/concentration-time curve from the time 0 to the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
h*IU/mL | 9.7836 (1.75225) | 8.7967 (1.64043)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Geometric least square mean ratio = 111.39, 95% CI 2-sided [105.89 to 117.17]

24. Secondary Outcome: AUC0-inf (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  AUC0-inf is the area under the activity/concentration-time curve from time 0 extrapolated to infinity. It was calculated as the sum of AUC0-t plus the ratio of the last measurable value to the elimination rate constant
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*IU/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 36 | 38
h*IU/mL | 9.1620 (1.47121) | 8.2160 (1.60673)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 10, analysis 1]; Geometric least square mean ratio = 113.82, 95% CI 2-sided [107.47 to 120.53]

25. Secondary Outcome: T1/2 (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  T1/2 is the apparent first-order terminal elimination half-life calculated as 0.693/kel.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 36 | 38
hours | 2.6595 (2.06574) | 1.9420 (1.47865)

26. Secondary Outcome: Cmin (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  Cmin is the minimun plasma activity/concentration.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: UI/mL
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 7 | 7
UI/mL | 0.000 (0.000) | 0.000 (0.000)

27. Secondary Outcome: Tmin (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  Tmin is the time of Cmin.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 9 | 12
hours | 0.00 (0.000) | 0.00 (0.000)

28. Secondary Outcome: AUC%ex (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  AUC%ex is the residual area, i.e. the percentage of the area under the curve (AUC) extrapolated to infinity observed from Tlast to infinity.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of total AUC
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 36 | 38
percentage of total AUC | 0.8078 (0.71131) | 0.6385 (0.52118)

29. Secondary Outcome: Tmax (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  Tmax is the time to Cmax.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 44 | 44
hours | 0.9973 (0.28432) | 0.9830 (0.24467)
Statistical Analysis 1: Comparison: Enoxaparin Sodium Chemi (Test IMP) vs Clexane (Reference IMP); Test type: Equivalence — [test comment as in outcome 17, analysis 1]; p = 0.9217, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0, 95% CI 2-sided [-0.13 to 0.13] — Median difference is the difference between median tmax in Test IMP versus Reference IMP arms

30. Secondary Outcome: Lambda Zeta (Anti-FXa/Anti-FIIa Ratio)
Description: The ratio of anti-FXa/anti-FIIa activity was calculated for each major parameter.
  Lambda zeta is the apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma activity/concentration vs time curve.
Time Frame: At day 1(0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h) and Day 2 (24 and 36h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Enoxaparin Sodium Chemi (Test IMP) | Clexane (Reference IMP)
Number analyzed (Participants) | 36 | 38
1/hour | 0.6699 (0.52191) | 1.0937 (1.82862)

ADVERSE EVENTS:
Time Frame: Throughout the study: day 1 (pre-dose,0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16h), Day 2 (24 and 36h), and post-study follow-up. Follow-up assessments were classified as 'End of study assessments'. They were performed on Day 2, 36 h post-dose, prior to discharging the subject.
Arm/Group | Enoxaparin Sodium Chemi | Clexane
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/45
Other Adverse Events (participants affected / at risk) | 7/46 | 5/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin Sodium Chemi (N=46) | Clexane (N=45)
Fibrous dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enoxaparin Sodium Chemi (N=46) | Clexane (N=45)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ligament sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No